CLINICAL TRIAL: NCT06810583
Title: A Prospective, Single-Arm, Trial of Dalbavancin-Based Prophylaxis in Children and Adolescents With High-Risk Leukemia
Brief Title: A Prospective Trial of Dalbavancin-Based Prophylaxis in Children and Adolescents With High-Risk Leukemia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAPHNE
Record Dates: First submitted 2025-01-06; First posted 2025-02-05 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Leukemia; Acute Myeloid Leukemia; Lymphoblastic Leukemia in Children
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute | interventions — dalbavancin; Fluoroquinolones

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- q28 days dalbavancin plus fluoroquinolone (Experimental): Dalbavancin given at standard treatment doses once every 28 days in combination with standard of care fluoroquinolone (ciprofloxacin or levofloxacin) prophylaxis.
  Interventions: Drug: Dalbavancin; Drug: Fluoroquinolone (either ciprofloxacin or levofloxacin at the discretion of the treating clinician)

INTERVENTIONS:
Drug: Dalbavancin — 3 doses of q28 days dalbavancin (12 weeks).
Drug: Fluoroquinolone (either ciprofloxacin or levofloxacin at the discretion of the treating clinician) — 28 days dalbavancin plus fluoroquinolone (either ciprofloxacin or levofloxacin at the discretion of the treating clinician) for up to 3 doses (12 weeks).

SUMMARY:
This is a single-arm pilot clinical trial evaluating dalbavancin-based prophylaxis in children and adolescents with acute myeloid leukemia or relapsed lymphoblastic leukemia receiving myelosuppressive chemotherapy.

Primary objective:

- To estimate the rate of bacterial bloodstream infection in pediatric patients with AML or relapsed ALL undergoing chemotherapy receiving dalbavancin-based prophylaxis

Secondary objectives:

* To describe the population pharmacokinetics of every 28 days dalbavancin up to 12 weeks in pediatric patients with AML or relapsed ALL undergoing chemotherapy
* To describe the tolerability of every 28 days dalbavancin prophylaxis in pediatric patients with AML or relapsed ALL undergoing chemotherapy
* To describe the acceptability of every 28 days dalbavancin prophylaxis in pediatric patients with AML or relapsed ALL undergoing chemotherapy
* To estimate the rates of likely bacterial infections, Clostridioides difficile infection, and febrile neutropenia in pediatric patients receiving dalbavancin-based prophylaxis

DETAILED DESCRIPTION:
Single-arm, open label, prospective, study with q28 days dalbavancin plus fluoroquinolone (either ciprofloxacin or levofloxacin at the discretion of the treating clinician) for up to 3 doses (12 weeks). Primary outcome will be rate of bacterial bloodstream infection during the first 56 days, with comparison to historical control receiving vancomycin-based prophylaxis (matched St. Jude cohort), or levofloxacin prophylaxis (published data Alexander et al, JAMA, 2018).

Participants will be enrolled, and consent obtained by experienced study staff. Baseline samples, including stool, will be collected within 72 hours after the first dose of dalbavancin. Participants will receive up to 3 doses of q28 days dalbavancin, plus ciprofloxacin or levofloxacin at the discretion of the treating clinician, until 12 weeks or other off study criteria are met. PK samples will be obtained after the first dose of dalbavancin and immediately prior to each subsequent dose. Participants will be monitored for adverse events related to dalbavancin, but adverse events directly related to leukemia or cancer therapy will not be reported.

ELIGIBILITY:
Inclusion Criteria:

* Aged less than or equal to 25 years at enrollment
* Receiving treatment for AML or relapsed ALL at St. Jude and treatment is expected to cause prolonged (> 7 days) severe neutropenia (ANC < 500/ml)
* Expected to receive care at St. Jude for at least 56 days following enrollment on the protocol
* Female participant, greater than or equal to 9 years old, has a documented negative pregnancy test prior to receipt of study drug.

Exclusion Criteria:

* Allergy to vancomycin, dalbavancin, teicoplanin, levofloxacin or ciprofloxacin (Not including non-anaphylactic vancomycin infusion reaction)
* Documented past or current infection or colonization with pathogenic bacteria resistant to vancomycin plus either ciprofloxacin or levofloxacin
* Diagnosed with long QT syndrome
* Any condition judged by the investigator to put the participant at high risk from participation
* Suspected or proven active bacterial infection
* Inability to complete requirements of participation in the study (in the opinion of the investigator)
* Expected survival <28 days
* Alkaline phosphatase, alanine transferase or total bilirubin ≥ 3x upper limit of normal for age
* Estimated glomerular filtration rate (EGFR) <30 mL/minute/1.73 m2
* Other absolute contraindication to administration of fluoroquinolone antibiotics or dalbavancin
* Participant is pregnant or breastfeeding a child

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 29 (Estimated)
Dates: Start 2025-05-22 (Actual); Primary Completion 2030-09 (Estimated); Study Completion 2031-09 (Estimated)

PRIMARY OUTCOMES:
Bacterial bloodstream infection | Day 56
  Proportion of evaluable participants with bacterial bloodstream infection with 95% confidence intervals

SECONDARY OUTCOMES:
Tolerability of dalbavancin | Day 56
  Proportion of evaluable participants with adverse events attributable to dalbavancin with 95% confidence intervals
Acceptability of dalbavancin prophylaxis | Day 56
  Median and range of TSQM II results
Likely bacterial infections, Clostridioides difficile infection, and febrile neutropenia | Day 84
  Proportion of evaluable participants with likely bacterial infections, Clostridioides difficile infection, or febrile neutropenia, with 95% confidence intervals
Dalbavancin peak plasma concentration (Cmax) - Median and range | Once
  Peak concentration of dalbavancin 30-60 minutes after completion of dose administration
Dalbavancin trough plasma concentration (Cmin)- Median and range | Up to 3 occasions over 87 days
  Trough concentration of dalbavancin 25-31 days after dose administration
Dalbavancin area under the concentration-time curve - Median and range | Once following first dose
  Estimated area under dalbavancin concentration-time curve

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Wolf, MBBS, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols